CLINICAL TRIAL: NCT05141721
Title: A Phase 2/3, Randomized, Open-Label Study of Maintenance GRT-C901/GRT-R902, A Neoantigen Vaccine, in Combination With Immune Checkpoint Blockade for Patients With Metastatic Colorectal Cancer
Brief Title: A Study of a Patient-Specific Neoantigen Vaccine in Combination With Immune Checkpoint Blockade for Patients With Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seattle Project Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO-010
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal cancer vaccine; mCRC; colon; rectum; CRC; rectal; immunotherapy; MSS-CRC; personal cancer vaccine; personalized cancer vaccine; individualized cancer vaccine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; Ipilimumab; Leucovorin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccine Arm (Experimental): After receiving up to 24 weeks induction therapy with a fluoropyrimidine/oxaliplatin/bevacizumab (with or without irinotecan), per standard of care and after completing vaccine production screening, patients will receive a total of 6 administrations of GRT-C901/GRT-R902 plus ipilimumab co-administered only with the first dose of GRT-C901 and GRT-R902. All patients will receive atezolizumab in addition to maintenance therapy of a fluoropyrimidine and bevacizumab according to standard of care.
  Interventions: Drug: GRT-C901; Drug: GRT-R902; Drug: Atezolizumab; Drug: Ipilimumab; Drug: Fluoropyrimidine plus leucovorin; Drug: Bevacizumab
- Control Arm (Active Comparator): After receiving up to 24 weeks induction therapy with a fluoropyrimidine/oxaliplatin/bevacizumab (with or without irinotecan), per standard of care and undergoing vaccine production screening, patients will receive maintenance therapy of a fluoropyrimidine and bevacizumab according to standard of care.
  Interventions: Drug: Fluoropyrimidine plus leucovorin; Drug: Bevacizumab

INTERVENTIONS:
Drug: GRT-C901 — A patient-specific neoantigen cancer vaccine administered via intramuscular (IM) injection as prime and single boost at a dose of 1x10^12 viral particles 2 times over the course of the first year.
  Arms: Vaccine Arm
Drug: GRT-R902 — A patient-specific neoantigen cancer vaccine boost, administered via IM injection at a dose of 30ug 4 times over the course of the first year.
  Arms: Vaccine Arm
Drug: Atezolizumab — Atezolizumab will be administered via intravenous (IV) infusion at a dose of 1680 mg once every 4 weeks.
  Other Names: Tecentriq
  Arms: Vaccine Arm
Drug: Ipilimumab — Ipilimumab will be administered via subcutaneous (SC) injection at a dose of 30 mg with the first dose of GRT-C901 and GRT-R902.
  Other Names: Yervoy
  Arms: Vaccine Arm
Drug: Fluoropyrimidine plus leucovorin — Fluoropyrimidine (infusional 5-FU or capecitabine) and leucovorin administered as maintenance therapy per standard of care.
  Other Names: Xeloda
Drug: Bevacizumab — Bevacizumab administered as maintenance therapy per standard of care.
  Other Names: Avastin

SUMMARY:
The primary objective of the Phase 2 portion of the study is to characterize the clinical activity of maintenance therapy with GRT-C901/GRT-R902 (patient-specific vaccines) in combination with checkpoint inhibitors in addition to fluoropyrimidine/bevacizumab versus a fluoropyrimidine/bevacizumab alone as assessed by molecular response which is based on changes in circulating tumor (ct)DNA. The primary objective of the Phase 3 portion is to demonstrate clinical efficacy of the regimen as assessed by progression-free survival.

DETAILED DESCRIPTION:
Tumors harboring non-synonymous deoxyribonucleic acid (DNA) mutations can present peptides containing these mutations as non-self antigens in the context of human leukocyte antigens (HLAs) on the tumor cell surface. A fraction of mutated peptides result in neoantigens capable of generating T-cell responses that exclusively target tumor cells. Sensitive detection of these mutations allows for the identification of neoantigens unique to each patient's tumor to be included in a patient-specific cancer vaccine that targets these neoantigens. This vaccine regimen uses two vaccine vectors as a heterologous prime/boost approach (GRT-C901 first followed by GRT-R902) to stimulate an immune response. This study will explore the anti-tumor activity of this patient-specific immunotherapy in combination with checkpoint inhibitors in addition to fluoropyrimidine/bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic colorectal cancer (CRC) who are planned for, or have received <30 days of first-line treatment in the metastatic setting with FOLFOX/bev, CAPEOX/bev, FOLFOXIRI/bev, or CAPOXIRI/bev per SOC
* Measurable and unresectable metastatic disease according to RECIST v1.1
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor specimens.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient has adequate organ function per defined criteria
* If women of childbearing potential (WCBP), must be willing to undergo pregnancy testing and agrees to the use at least 1 highly effective contraceptive method during the study treatment period and for 150 days after last investigational study treatment.

Exclusion Criteria:

* Patients with deficient mismatch repair (dMMR) or microsatellite instability (MSI-H) phenotype
* Patient has a known tumor mutation burden <1 non-synonymous mutations/megabase
* Known DNA Polymerase Epsilon mutations
* Patients with known BRAFV600E mutations
* Bleeding disorder or history of significant bruising or bleeding following IM injections or blood draws
* Immunosuppression anticipated at time of study treatment
* History of allogeneic tissue/solid organ transplant
* Active or history of autoimmune disease or immune deficiency
* Patient with symptomatic or actively progressing central nervous system (CNS) metastases, carcinomatous meningitis, or has been treated with whole brain radiation
* History of other cancer within 2 years with the exception of neoplasm that has undergone potentially curative therapy
* Any severe concurrent non-cancer disease that, in the judgment of the Investigator, would make the patient inappropriate for the current study
* Active tuberculosis or recent (<2 weeks) clinically significant infection, evidence of active hepatitis B or hepatitis C, or known history of positive test for HIV
* History of pneumonitis requiring systemic steroids for treatment (with the exception of prior resolved in-field radiation pneumonitis)
* Myocardial infarction within previous 3 months, unstable angina, serious uncontrolled cardiac arrhythmia, history of myocarditis, or congestive heart failure (Class III or IV).
* Pregnant, planning to become pregnant, or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-02-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Molecular response defined as ≥ 30% decrease from baseline in circulating tumor DNA (ctDNA) | Baseline and up to 27 months
Phase 3: Progression-free survival per Immune-based Response Evaluation Criteria in Solid Tumors (iRECIST) as assessed by blinded independent review committee (IRC) | Up to 60 months
  defined by time from randomization until disease progression as per iRECIST or death from any cause

SECONDARY OUTCOMES:
Phase 2 and 3: Incidence of treatment-emergent adverse events (TEAEs), immune-related AEs, treatment-related AEs, serious AEs, AEs leading to death, AEs leading to dose delays, and AEs leading to discontinuation of study treatment | Phase 2 up to 27 months, Phase 3 up to 60 months
Phase 2 and 3: Progression-free survival per RECIST v1.1 and iRECIST as assessed by the investigator | Phase 2: up to 27 months, Phase 3: up to 60 months
Phase 3: Progression-free survival per RECIST v1.1 as assessed by blinded IRC | Up to 60 months
Phase 2 and 3: Overall Survival as time from randomization to death from any cause | Phase 2 up to 27 months, Phase 3 up to 60 months
Phase 2 and 3: Overall Response Rate | Phase 2 up to 27 months, Phase 3 up to 60 months
  measured by the proportion of patients with best overall response (BOR) of partial response (PR) or complete response (CR) by REICST v1.1 or , immune-based PR (iPR) or immune-based by iRECIST
Phase 2 and 3: Duration of response (DOR) defined by time from the first objective response of PR or PR until disease progression or death | Phase 2 up to 27 months, Phase 3 up to 60 months
Phase 2 and 3: Clinical benefit rate (CBR) as defined by the proportion of patients with best overall response of stable disease (SD), PR or CR using RECIS v1.1 or immune-based SD (iSD), iPR, or iCR by iRECIST. | Phase 2 up to 27 months, Phase 3 up to 60 months
Phase 2 and 3: Deepening of Response the proportion of patients who have a BOR of SD or PR during the VPS and who convert from SD to PR or CR, or from PR to CR after start of the study treatment and/or SOC maintenance treatment in the STS per RECIST v1.1 | Phase 2 up to 27 months, Phase 3 up to 60 months
  VPS = Vaccine Production Stage; STS = Study Treatment Stage
Phase 2 and 3: The feasibility of manufacturing a patient-specific vaccine defined by the proportion of patients for whom vaccine was successfully manufactured from those randomized to the vaccine arm. | Study Treatment Screening visit (up to 28 days before Day 1 of study drug administration)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Banner MD Anderson, Gilbert, Arizona
  - Highlands Oncology, Springdale, Arkansas
  - U.S.C Norris Cancer Center, Keck School of Medicine, Division of Medical Oncology, Los Angeles, California
  - University of California - Irvine (UCI), Orange, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Rocky Mountain Cancer Centers - USOR, Denver, Colorado
  - Eastern CT Hematology and Oncology Associates (ECHO), Norwich, Connecticut
  - Lynn Cancer Institute - Boca Raton Regional Hospital, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - Miami Cancer Institute at Baptist Health South Florida (USOR site), Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Orlando Health, Orlando, Florida
  - Advanced Research (Oncology & Hemotology Associates of West Broward), Tamarac, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Fairway, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Astera Cancer Care, East Brunswick, New Jersey
  - Summit Health, Florham Park, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers, New Brunswick, New Jersey
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - New York Cancer and Blood, Port Jefferson Station, New York
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Northwest Cancer Specialists DBA Compass Oncology - USOR, Portland, Oregon
  - Sidney Kimmel Medical College at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Tennessee Oncology - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology PA - USOR, Austin, Texas
  - Texas Oncology - Dallas Sammons, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Baylor Scott and White, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No